CLINICAL TRIAL: NCT02451098
Title: A Multicenter, Randomized, Double-blind, Active-controlled, Parallel Group, Factorial Design, Phase III Clinical Trial To Evaluate the Efficacy and Safety of Atorvastatin+Ezetimibe Combination Therapy and Atorvastatin Monotherapy in Patients With Primary Hypercholesterolemia
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of CKD-391
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 152PDL14025
Record Dates: First submitted 2015-05-18; First posted 2015-05-21 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Atorvastatin10mg, Ezetimibe10mg (Experimental): Atorvastatin10mg, Ezetimibe10mg will be administered (Duration 8 weeks)
  Interventions: Drug: Atorvastatin10mg, Ezetimibe10mg
- Atorvastatin10mg, Ezetimibe placebo (Active Comparator): Atorvastatin10mg, placebo will be administered (Duration 8 weeks)
  Interventions: Drug: Atorvastatin10mg, Ezetimibe placebo
- Atorvastatin20mg, Ezetimibe10mg (Experimental): Atorvastatin20mg, Ezetimibe10mg will be administered (Duration 8 weeks)
  Interventions: Drug: Atorvastatin20mg, Ezetimibe10mg
- Atorvastatin20mg, Ezetimibe placebo (Active Comparator): Atorvastatin20mg, placebo will be administered (Duration 8 weeks)
  Interventions: Drug: Atorvastatin20mg, Ezetimibe placebo
- Atorvastatin40mg, Ezetimibe10mg (Experimental): Atorvastatin40mg, Ezetimibe10mg will be administered (Duration 8 weeks)
  Interventions: Drug: Atorvastatin40mg, Ezetimibe10mg
- Atorvastatin40mg, Ezetimibe placebo (Active Comparator): Atorvastatin40mg, placebo will be administered (Duration 8 weeks)
  Interventions: Drug: Atorvastatin40mg, Ezetimibe placebo

INTERVENTIONS:
Drug: Atorvastatin10mg, Ezetimibe10mg — Atorvastatin10mg, Ezetimibe 10mg (Duration: 8weeks)
  Other Names: CKD-391
  Arms: Atorvastatin10mg, Ezetimibe10mg
Drug: Atorvastatin10mg, Ezetimibe placebo — Atorvastatin10mg, Ezetimibe placebo(Duration: 8 weeks)
  Other Names: Lipitor
  Arms: Atorvastatin10mg, Ezetimibe placebo
Drug: Atorvastatin20mg, Ezetimibe10mg — Atorvastatin20mg, Ezetimibe 10mg (Duration: 8weeks)
  Other Names: CKD-391
  Arms: Atorvastatin20mg, Ezetimibe10mg
Drug: Atorvastatin20mg, Ezetimibe placebo — Atorvastatin20mg, Ezetimibe placebo(Duration: 8weeks)
  Other Names: Lipitor
  Arms: Atorvastatin20mg, Ezetimibe placebo
Drug: Atorvastatin40mg, Ezetimibe10mg — Atorvastatin40mg, Ezetimibe 10mg (Duration: 8weeks)
  Other Names: CKD-391
  Arms: Atorvastatin40mg, Ezetimibe10mg
Drug: Atorvastatin40mg, Ezetimibe placebo — Atorvastatin40mg, Ezetimibe placebo(Duration: 8weeks)
  Other Names: Lipitor
  Arms: Atorvastatin40mg, Ezetimibe placebo

SUMMARY:
A Multicenter, Randomized, Double-blind, Active-controlled, Parallel group, Factorial Design, Phase III Clinical Trial.

DETAILED DESCRIPTION:
The aim of this phase 3 study was to evaluate the efficacy and safety of CKD-391 once daily for 8 weeks in patients with primary hypercholesterolemia. Furthermore, the extension study for additional 12 weeks is designed to confirm long term safety of CKD-391.

ELIGIBILITY:
Inclusion Criteria:

* Adult, at least 19 years of age.
* Hyperlipidemia patient of LDL-C≤250 mg/dl and TG ≤400 mg/dl
* Patients requiring anti-dyslipidemia drug therapy [based on the NCEP ATP III(2002)]
* Drug compliance during Run-in period ≥70%
* Patients must willing to the study and signed an informed consent

Exclusion Criteria:

* Patients with myopathy included rhabdomyolysis or CPK level≥2xULN
* Patients with acute arterial disease
* Patients with renal dysfunction or Serum creatinine level ≥2x ULN
* Patients with liver dysfunction or ALT, AST level > 2xULN
* Patients with medical history within 6 months prior to screening visit (Heart failure, uncontrolled arrhythmia, drug and alcohol abuse history, gastrointestinal disease or surgery, anticoagulation disease)
* Patient with uncontrolled disease (diabetes mellitus as HbA1c level of > 9.0%, hypertension as SBP≥180mmHg or DBP≥110mmHg, hypothyroidism as TSH≥1.5xULN)
* Patients who have a history or presence of active malignancy within 5 years
* Patients with difficulty of stop taking lipid-lowering agents during run-in period.
* Patients who have taken another investigational drug within 4 weeks prior to screening visit.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change form baseline in LDL-C | up to week 8

SECONDARY OUTCOMES:
Change form baseline in LDL-C | up to week 20
Change form baseline in Total cholesterol | up to week 20
Change form baseline in Triglyceride | up to week 20
Change form baseline in HDL-C | up to week 20
Change form baseline in Non-HDL-C | up to week 20
Change form baseline in LDL-C/HDL-C ratio | up to week 20
Change form baseline in TC/HDL-C ratio | up to week 20
Change form baseline in Non-HDL-C/HDL-C ratio | up to week 20
Change form baseline in Apo-B ratio | up to week 20
Change form baseline in Apo-B | up to week 20
Change form baseline in Apo-A1 | up to week 20
Change form baseline in Apo-B/Apo-A1 ratio | up to week 20

OTHER OUTCOMES:
Evaluate safety of CKD-391 from adverse events, laboratory test results, physical examination, vital signs. | up to week 20

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Jung Yoon, PhD, Principal Investigator — The Catholic University of Korea
Locations (1):
- The catholic university of korea seoul st. Mary's hospital, Seoul, South Korea